CLINICAL TRIAL: NCT00455897
Title: Phase II Trial of CHOP-Rituximab Augmented With Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in Patients With Previously Untreated Diffuse Large B Cell Non-Hodgkin's Lymphoma
Brief Title: CHOP-Rituximab Augmented With GM-CSF in Patients With Previously Untreated Diffuse Large B Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual was too slow. Trial terminated
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); Bayer (Industry)
Responsible Party: Principal Investigator, Ephraim Hochberg, MD, Director Clinical Lymphoma Research, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-342
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Diffuse
Keywords: granulocyte monocyte colony stimulating factor; Leukine; Sargramostim; Diffuse large B cell lymphoma; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GMCSF-RCHOP (Experimental)
  Interventions: Drug: GM-CSF; Drug: CHOP; Drug: Rituximab

INTERVENTIONS:
Drug: GM-CSF — Given 11 days before day 1 of cycle 1 for 10 days
Drug: CHOP — Administered as part of standard care
Drug: Rituximab — Administered as part of standard treatment

SUMMARY:
The primary goal of this study is to determine the effects (good and bad) of Granulocyte-macrophage colony stimulating factor (GM-CSF) in combination with Cytoxan, Adriamycin, Vincristine, Prednisone, Rituximab (CHOP-R) on diffuse Large B cell Non-Hodgkin's lymphoma (DLBCL). The standard of care for DLBCL is the combination of drugs known as CHOP-Rituximab (CHOP-R). The drugs that make up CHOP-R are the chemotherapy drugs cyclophosphamide, doxorubicin and vincristine, prednisone and rituximab. GM-CSF is a drug that stimulates the immune system by increasing the numbers of white blood cells. Previous research has shown that GM-CSF might help rituximab to be more effective in treating lymphoma.

DETAILED DESCRIPTION:
* Study treatment is divided into 21-day time periods called cycles. Almost all participants will be treated as outpatients unless they have an existing medical problem that requires them to be treated as in inpatient.
* The drugs used in this study treatment are standard of care for this type of lymphoma and participants could receive these even if they are not taking part in the study.
* Participants will start receiving GM-CSF 11 days before Day 1 of Cycle 1 for 10 days. They will receive the first dose of GM-CSF at the clinic. At least 1 1/2 days after the last GM-CSF injection (Day 1), they will receive chemotherapy (CHOP-R). Eleven days before they start the next cycle (Days 11-20), they will again start to receive GM-CSF injections for 10 days.
* Participants will receive up to 6 cycles of study treatment if their disease is responding and they are tolerating the study treatment.
* Additional medications may be given to prevent lung infection, return of brain and nervous system disease and tumor lysis syndrome.
* Before beginning GM-CSF during each cycle of treatment blood will be drawn to monitor the participants health and to check for side effects.
* On Day 1 of each cycle a physical examination and blood tests will be performed. On Day 7 and Day 14 of each cycle, routine blood tests will also be done.
* After Cycle 2 and 4 CT scans of the neck, chest, abdomen and pelvis will be performed to check the status of the participants disease.
* After 6 cycles of study treatment, the participant will return to the clinic for an End of Treatment Visit. At this visit a physical exam, routine blood tests, and CT scan of neck, chest, abdomen and pelvis will be performed.
* The participant will be asked to return to the clinic every 3 months for the first year after study treatment and every 6 months up to 2 years after study treatment for the procedures outline in the End of Treatment Visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of diffuse large B cell Non-Hodgkin's lymphoma with characteristic immunophenotypic profile
* Patient has not received any prior anti-cancer therapy for lymphoma
* Tumor tissue confirmed to express the cluster of differentiation antigen 20 antigen by flow cytometry or immunohistochemistry
* Measurable disease as defined by a tumor mass of 1cm or greater in one dimension
* Stage II (abdominal-not radiotherapy appropriate), III, or IV disease
* Age > 18 years
* Performance Status of 0-2
* Laboratory parameters as outlined in protocol
* Patient agrees to use birth control

Exclusion Criteria:

* Known central nervous system involvement by lymphoma
* Serious uncontrolled concurrent illness such as active coronary artery disease, severe lung disease, heart failure, active alcohol abuse, active concurrent malignancy except non-melanoma skin cancer or carcinoma in situ of the cervix
* Any evidence of prior natural exposure to Hepatitis B
* Active rheumatologic disease which may be exacerbated by GM-CSF
* Cardiac ejection fraction less than 45%
* Known HIV disease
* Patient is pregnant or nursing
* Patient is receiving other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety of GM-CSF when administered in combination with CHOP-R to patients with previously untreated diffuse large B cell non-Hodgkin's lymphoma. | 2 years

SECONDARY OUTCOMES:
To assess the response rate, 2-year event-free survival and overall survival with CM-CSF and CHOP-R in this patient population
to analyze the biologic activity of GM-CSF at this dosing schedule and timing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim P Hochberg, MD, Principal Investigator — Massachusetts General Hosptial
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts